CLINICAL TRIAL: NCT02387333
Title: Role of Mesh Stoma Reinforcement Technique (MSRT) in Prevention of Parastomal Hernia After Ileal Conduit Urinary Diversion: A Randomized Controlled Trial
Brief Title: Role of Mesh Stoma Reinforcement Technique (MSRT) in Prevention of Parastomal Hernia After Ileal Conduit Urinary Diversion
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Amr Abdel-Lateif El-Sawy, Resident in Urology, Urology and Nephrology Center, Mansoura University, Mansoura, Egypt, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AEl-Sawy132015
Record Dates: First submitted 2015-02-28; First posted 2015-03-13 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Ileal Conduit; Parastomal Hernia
Keywords: Radical cystectomy; Urinary diversion; Ileal conduit; Parastomal hernia; Prophylactic mesh; Mesh stoma reinforcement technique
MeSH Terms: interventions — Urinary Diversion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study group (Experimental): in this arm -study group- : patients will receive mesh stoma reinforcement technique with ileal conduit urinary diversion.
  Interventions: Procedure: Polypropylene Mesh Stoma reinforcement technique with ileal conduit urinary diversion
- Control group (Sham Comparator): in this arm -sham comparator- : patients will not receive mesh stoma reinforcement technique with ileal conduit urinary diversion.
  Interventions: Procedure: Ileal conduit urinary diversion

INTERVENTIONS:
Procedure: Polypropylene Mesh Stoma reinforcement technique with ileal conduit urinary diversion — After standard steps of radical cystectomy and sparing of distal 15 cm of ileum as a conduit for diversion.
  A preferred rectal muscle splitting approach is preferred for IC exteriorization.
  Dissection of subcutaneous fat off the rectus sheath will be accomplished to create a potential space for mesh placement.
  Then, 5 x 5 cm polypropylene mesh will be placed and incised at the center to create an orifice to allow IC exteriorization.
  The mesh is then fixed to underlying rectus sheath with 1-0 non-absorbable proline sutures.
  The IC is exteriorized through the central orifice and then fixed to the peritoneum and to the cut-edges of the rectus muscle using 3-0 polyglactin sutures.
  A 12 CH subcutaneous tube drain will be left and the subcutaneous tissue is closed to collapse the dissected space around the mesh.
  The stoma is then everted and fixed to the skin.
  Other Names: Implantable polypropylene monofilament mesh
  Arms: Study group
Procedure: Ileal conduit urinary diversion — In this group, no mesh will be applied with ileal conduit urinary diversion
  Arms: Control group

SUMMARY:
The aim of this clinical trial is to investigate the safety and efficacy of prophylactic mesh on prevention of parastomal hernia(PSH) after ileal conduit urinary diversion (IC) in a randomized controlled fashion.

DETAILED DESCRIPTION:
All patients will be recruited from the urology practice of the study's investigators, Urology department of Urology and Nephrology Center (UNC), Mansoura university, Egypt. Patients will be asked to participate after the patient and physician have made a decision that ileal conduit urinary diversion of choice. Those patients meeting all inclusion criteria will be asked to participate in this study with informed consent then obtained. No monetary income will be offered for participation in the study.

Those patients will be evaluated clinically and radiologically according to the specified protocol.

After enrollment in the study, the stoma site will be marked on the skin the day prior to surgery by the stoma therapist. All patients will be operated by high volume surgeon experienced in IC urinary diversion. The procedure started by radical cystectomy and bilateral pelvic lymphadenectomy. After sparing the distal 15 cm of the terminal ileum, a 15 cm ileal segment will be isolated and the bowel continuity will be restored and the mesenteric defect will be closed. The distal end of the isolated bowel segment will be mobilized and exteriorized at the predetermined site on the abdominal wall followed by stoma eversion. A preferred rectal muscle splitting approach is preferred for IC exteriorization. In case of MSRT, dissection of subcutaneous fat off the rectus sheath will be accomplished to create a potential space for mesh placement. Then, 5 x 5 cm polypropylene mesh will be placed and incised at the center to create an orifice to allow IC exteriorization. The mesh is then fixed to underlying rectus sheath with 1-0 non-absorbable proline sutures. The IC is exteriorized through the central orifice and then fixed to the peritoneum and to the cut-edges of the rectus muscle using 3-0 polyglactin sutures. A 12 CH subcutaneous tube drain will be fixed and the subcutaneous tissue is closed to collapse the dissected space around the mesh. The stoma is then everted and fixed to the skin. Sham group patients will undergo the same technique without mesh placement. The ureters will be mobilized and anastomosed to the proximal end of the conduit using direct ureteroileal anastomosis.

All patients will undergo the routine protocol at the investigators' center including enrollment in fast track restoration of bowel habits, ileal conduit catheter to be removed on the 5th day and the ureteral stents on the 7th and 8th days. Any deviation from normal postoperative course will be recorded using the modified Clavien-Dindo system.

At followup, patients will be asked to attend the outpatient clinic at 1, 3, 6, and 12 months after discharge clinically and radiologically to assess the intended outcomes of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to give informed consent.
2. Patients with history of chronic liver disease
3. Patients with history of systemic chemotherapy, radiotherapy or maintenance on systemic corticosteroids
4. Patients with chronic causes of increased intra-abdominal pressure as chronic cough (COPD) or chronic constipation
5. Patients with surgical history of hernia repair
6. Patients with body mass index (BMI) more than 30 kg/m2
7. Patients with other hernias (inguinal, umbilical or incisional) at preoperative evaluation
8. Patients with low serum albumin < 3 gm/dl
9. Patients who will be highly candidates for adjuvant or palliative chemo-radiotherapy such those with histopathologically proved residual tumor

Exclusion Criteria:

1. Inability to give informed consent.
2. Patients who documented previous allergic reaction to synthetic mesh.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-02; Primary Completion 2018-10 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of parastomal hernia 2 years after surgery | 2 years
  The primary outcome of this study will be the incidence of parastomal hernia at 2 years after surgery

SECONDARY OUTCOMES:
Adverse events related to mesh placement | 2 years
  The secondary outcome will be the adverse events related to mesh placement.
Health related quality of life as measured by Body Image Scale (BIS) questionnaire | 2 years
  Health related quality of life issues will be assessed also in both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed E. Mosbah, MD, Study Chair — Urology And Nephrology Center, Mansoura University, Mansoura
Locations (1):
- Urology and Nephrology Center, Al Mansurah, DK, Egypt